CLINICAL TRIAL: NCT05359211
Title: A Phase Ib Open-Label Study Evaluating the Safety and Efficacy of NKTR-255 in Combination With CD19-Directed CAR-T Cell Therapy in Patients With Relapsed/Refractory (R/R) Large B-Cell Lymphoma (LBCL)
Brief Title: NKTR-255 in Combination With CAR-T Cell Therapy for the Treatment of Relapsed or Refractory Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1122036; NCI-2022-02316 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10802 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Grade 3b Follicular Lymphoma; Recurrent Primary Mediastinal Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory Grade 3b Follicular Lymphoma; Refractory Primary Mediastinal Large B-Cell Lymphoma; Transformed Indolent B-Cell Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; fludarabine; NKTR-255; X-Rays; Phantoms, Imaging; Spinal Puncture; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lymphodepletion, liso-cel, NKTR-255) (Experimental): Patients receive standard of care lymphodepletion therapy consisting of cyclophosphamide and fludarabine on days -5 to -3 followed by liso-cel CAR-T cell infusion on day 0. Patients then receive NKTR-255 IV over 30 minutes every 3 weeks starting on day 10 or 14 for up to 3 doses in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray and ECHO or MUGA during screening. Patients undergo bone marrow biopsy and aspiration, LP for CSF sample collection during screening, on the study and during follow-up as clinically indicated. Patients also undergo PET/CT throughout the trial. Additionally, patients undergo blood sample collection and may optionally undergo tissue biopsy throughout the trial.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Lisocabtagene Maraleucel; Drug: Polymer-conjugated IL-15 Receptor Agonist NKTR-255; Procedure: X-Ray Imaging; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Lumbar Puncture; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Biospecimen Collection; Procedure: Biopsy

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; Asta B 518; B-518
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Lisocabtagene Maraleucel — Given IV
  Other Names: Anti-CD19-CAR Genetically Engineered Autologous T Lymphocytes JCAR017; Anti-CD19-CAR Genetically Engineered Autologous T-lymphocytes JCAR017; Autologous Anti-CD19-EGFRt-4-1BB-zeta-modified CAR CD8+ and CD4+ T-lymphocytes JCAR017; Breyanzi; JCAR 017; JCAR017; Liso-cel
Drug: Polymer-conjugated IL-15 Receptor Agonist NKTR-255 — Given IV
  Other Names: IL-15 Receptor Agonist NKTR-255; Long-acting Polymer-conjugated IL-15; NKTR 255; NKTR-255; NKTR255
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging; Plain film radiographs; Radiographic Imaging
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Synchronized Multigated Acquisition Scanning; RNVG; SYMA Scanning
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; spinal tap
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT Scan; Computed Axial Tomography; CT; CT SCAN
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging; PET; PET scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: Bx

SUMMARY:
This phase Ib trial studies the effects of NKTR-255 in combination with chimeric antigen (CAR)-T cell therapy and to see how well they work in treating patients with large B-cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). NKTR-255 is an investigational IL-15 receptor agonist designed to boost the immune system's natural ability to fight cancer. T cells are infection fighting blood cells that can kill tumor cells. Lisocabtagene maraleucel is a CAR-T cell product that consists of genetically engineered T cells, modified to recognize CD19, a protein on the surface of cancer cells. These CD19-specific T cells may help the body's immune system identify and kill CD19-positive cancer cells. Giving NKTR-255 together with lisocabtagene maraleucel may work better in treating large B-cell lymphoma than either drug alone.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive standard of care lymphodepletion therapy consisting of cyclophosphamide and fludarabine on days -5 to -3 followed by liso-cel CAR-T cell infusion on day 0. Patients then receive NKTR-255 intravenously (IV) over 30 minutes every 3 weeks starting on day 10 or 14 in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray and echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients undergo bone marrow biopsy and aspiration, lumbar puncture (LP) for cerebrospinal fluid (CSF) sample collection during screening, on the study and during follow-up as clinically indicated. Patients also undergo positron emission tomography (PET)/computed tomography (CT) throughout the trial. Additionally, patients undergo blood sample collection and may optionally undergo tissue biopsy throughout the trial.

After completion of study treatment, patients are followed up every 30 days then every 3 months up to 12 months after the CAR-T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age at the time of consent
* Patients with LBCL (including diffuse large B-cell lymphoma [DLBCL] not otherwise specified [including DLBCL arising from indolent lymphoma], high-grade B-cell lymphoma, primary mediastinal large B-cell lymphoma, and follicular lymphoma grade 3B) with a Food and Drug Administration (FDA)-approved indication for treatment with liso-cel
* Fludeoxyglucose F-18 (FDG)-avid disease on positron emission tomography (PET) imaging or pathology evidence of active disease
* Evidence of CD19 expression on any prior or current tumor specimen or a high likelihood of CD19 expression based on disease histology
* Karnofsky performance status >= 60%
* Absolute neutrophil count (ANC) >= 1000 cells/mm^3 in the absence of bone marrow involvement by lymphoma
* Platelets >= 50,000 cells/mm^3 in the absence of bone marrow involvement by lymphoma
* Hemoglobin >= 8 g/dL in the absence of bone marrow involvement by lymphoma
* Calculated creatinine clearance (Cockcroft/Gault) > 30 mL/min/1.73 m^2
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (or < 5 x ULN for subjects with lymphomatous infiltration of the liver)
* Total bilirubin =< 2 (or < 3.0 for subjects with Gilbert's syndrome or lymphomatous infiltration of the liver)
* Common Terminology Criteria for Adverse Events (CTCAE) Grade =< 1 dyspnea
* Saturation of oxygen (Sa02) >= 92% on room air
* Patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing and must have a forced expiratory volume in 1 second (FEV1) of >= 50% of predicted value
* Patients with clinically significant pulmonary dysfunction, as determined by medical history and physical exam should undergo pulmonary function testing and must have a diffusing capacity of the lung for carbon monoxide (DLCO; corrected) >= 40% of predicted value
* Left ventricular ejection fraction (LVEF) >= 40% as assessed by echocardiogram or multiple uptake gated acquisition (MUGA)
* Patients with Fridericia's corrected QT interval (QTcF) > 450 ms for men and > 470 ms for women will require clearance by a cardiologist
* Women of reproductive potential (defined as all women physiologically capable of becoming pregnant) must agree to use suitable methods of contraception for 1 month after the last dose of study therapy (NKTR-255)
* Males who have partners of reproductive potential must agree to use an effective barrier contraceptive method for 1 month after the last dose of study therapy (NKTR-255)
* Ability to understand and provide informed consent
* Able and willing to comply with study visit schedule and procedures, including tumor biopsy where feasible and with acceptable risk

Exclusion Criteria:

* Planned use of therapeutic doses of corticosteroids (> 20 mg/day prednisone or equivalent) or other systemic immunosuppression within 7 days prior to leukapheresis or within 72 hours prior to liso-cel infusion. Topical and/or inhaled steroids are permitted
* Prior treatment with any CD19 CAR-T cell therapy
* For allogeneic hematopoietic cell transplant (HCT) recipients, active graft versus host disease (GVHD) and/or systemic GVHD therapy within 30 days prior to planned leukapheresis
* Known active hepatitis B (detectable hepatitis B deoxyribonucleic acid [DNA]) or hepatitis C (detectable hepatitis C ribonucleic acid [RNA])
* Known human immunodeficiency virus (HIV) infection
* Pregnant or breastfeeding women
* Prior treatment with any IL-2 or IL-15 agonist and/or biosimilar agents
* Active autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., ulcerative colitis, Crohn's disease], celiac disease, or other serious chronic gastrointestinal conditions associated with diarrhea, autoimmune vasculitis, systemic lupus erythematosus, Wegener syndrome [granulomatosis with polyangiitis], myasthenia gravis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.) requiring immunosuppressive therapy. The following are exceptions to this criterion:

  * Vitiligo.
  * Alopecia.
  * Hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
  * Type 1 diabetes mellitus.
  * Psoriasis not requiring systemic treatment.
  * Conditions considered to be low risk of serious deterioration by the principal investigator (PI).
* History of any one of the following cardiovascular conditions within the past 6 months: class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, or unstable angina; unless clearance by a cardiologist is obtained. History of other clinically significant cardiac disease that, in the opinion of the PI or designee, is a contraindication to study treatment is also excluded
* History or presence of clinically relevant central nervous system (CNS) pathology, such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, or psychosis that in the opinion of the PI is a contraindication to study treatment.

  * Patients with active parenchymal CNS involvement by malignancy will be excluded. Patients with prior or current secondary leptomeningeal CNS disease are eligible. CNS disease prophylaxis must be stopped at least 1 week prior to liso-cel infusion
* History of solid organ transplantation
* Active, serious, and uncontrolled infection(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 30 days after the last dose of NKTR-255 or until a new antitumor therapy has been initiated
  Grade ≥ 3 AEs considered related to NKTR-255 will be listed and summarized. Summaries of grade ≥ 3 laboratory data will include, at a minimum, treatment-emergent laboratory abnormalities. Summaries of AEs and laboratory abnormalities will be based on the safety evaluable population.
Dose-limiting toxicity (DLT) rates | Up to 21 days after the first NKTR-255 infusion
  Observed DLT rates will be summarized based on the DLT evaluable population. Final DLT rates at each dose level will be estimated by isotonic regression by applying the pooled adjacent violators algorithm.
Optimal biological dose (OBD) | Up to 12 months after the CAR-T cell infusion
  A composite of clinical information will be utilized to determine the OBD based on safety and tolerability, confirmation of maximum target engagement, optimal biological effects without undesirable clinical effects, pharmacokinetic parameters, and biological response data.
Complete response (CR) rate | Up to 3 months after the CAR-T cell infusion
  The CR rate will be summarized along with the 2-sided 95% exact Clopper-Pearson confidence interval based on the efficacy evaluable population.

SECONDARY OUTCOMES:
Complete response (CR) and overall response (OR) rates | Up to 12 months after the CAR-T cell infusion
  The CR and OR rates will be summarized along with the 2-sided 95% exact Clopper-Pearson confidence interval based on the efficacy evaluable population.
Duration of response (DOR) | Up to 12 months after the CAR-T cell infusion
  Will be assessed among responders. If a patient does not have an event for the DOR analyses, the patient will be censored at the date of the last adequate disease assessments or prior to the earliest censoring event. The censoring reason can include last contact/follow-up, discontinuation or completion of the study, receipt of another anticancer treatment with the exception of consolidation therapy with hematopoietic cell transplantation (HCT), and at least two consecutive missed scheduled disease assessments. Kaplan-Meier (KM) method will be used to analyze DOR.
Progression free survival (PFS) | Up to 12 months after the CAR-T cell infusion
  Will be assessed among responders. If a patient does not have an event for the PFS analyses, the patient will be censored at the date of the last adequate disease assessments or prior to the earliest censoring event. The censoring reason can include last contact/follow-up, discontinuation or completion of the study, receipt of another anticancer treatment with the exception of consolidation therapy with HCT, and at least two consecutive missed scheduled disease assessments. KM method will be used to analyze PFS.
Overall survival (OS) | Up to 12 months after the CAR-T cell infusion
  Analyses of OS will be performed in the safety population. For assessment of OS, data from surviving patients will be censored at the last time that the patient is known to be alive. KM method will be used to analyze OS.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Hirayama, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT05359211/ICF_000.pdf